CLINICAL TRIAL: NCT00001133
Title: A Phase I/II, Randomized, Open-Label Study of the Safety and Pharmacokinetics of Indinavir + Ritonavir Therapy in HIV-Infected Subjects Failing Amprenavir, Nelfinavir, Saquinavir, or Nelfinavir/Saquinavir Combination Therapy
Brief Title: Safety and Tolerance of Indinavir Plus Ritonavir in HIV-Positive Patients Failing Therapy With Amprenavir, Nelfinavir, or Saquinavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5055; 10672 (Registry Identifier: DAIDS ES); ACTG A5055; AACTG A5055
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Indinavir; Anti-HIV Agents; Pharmacokinetics; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir

SUMMARY:
In this study, the protease inhibitors indinavir (IDV) and ritonavir (RTV) will be studied in patients who have high levels of virus while taking other protease inhibitors. The purpose of this study is to see how the body takes in, distributes, and gets rid of IDV and RTV. This study will also look at any side effects that IDV or RTV causes.

IDV is an effective anti-HIV drug, but it can be difficult for patients to take. For IDV to work against HIV, it must be taken 3 times a day at a high dose and with a certain diet. Doctors believe IDV may be easier to take if it is given with RTV. Patients who take IDV and RTV together may be able to take IDV only twice a day and at a lower dose. This study will gather information about the safety and side effects of using IDV and RTV together.

DETAILED DESCRIPTION:
IDV, a protease inhibitor, has shown excellent clinical and virologic responses when combined with 2 nucleoside analogues. Although effective, the pharmacokinetics of IDV make it difficult to use in many patients. The drug has a short half-life and requires administration in high doses every 8 hours with significant dietary restrictions. Research has shown that IDV kinetics can be improved significantly by the addition of RTV, allowing for administration of IDV at lower doses every 12 hours. The half-life of IDV is prolonged 3- to 5-fold when administered with RTV. Based on these results, it is reasonable to study this combination as a twice-daily dosing regimen.

Patients are randomized to receive 1 of 2 doses of IDV/RTV for 24 weeks (Arms A and B). All patients also receive 2 nucleoside reverse transcriptase inhibitors (NRTIs). The NRTIs are not provided by the study. Clinical assessments take place at Weeks 1, 2, 4, 8, 12, 16, 20, and 24 which includes a virology assessment. [AS PER AMENDMENT 4/21/00: Patients who experience a confirmed virologic failure (defined in protocol) and elect to remain on study treatment, are followed through Week 24. Patients who experience a confirmed virologic failure and elect to discontinue study treatment will have a final evaluation at the time of treatment discontinuation.] Patients are hospitalized for 12 hours at the Week 2 study visit for an intensive pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 18 years old.
* Have a viral load (level of HIV in the blood) of at least 500 copies/ml but no more than 100,000 copies/ml within 45 days of study entry.
* Have been taking the following anti-HIV drug combination for at least 12 weeks before study entry: 2 NRTIs plus amprenavir (APV), nelfinavir (NFV), saquinavir (SQV), or NFV plus SQV.
* Are naive to at least 1 NRTI. This means that there is at least 1 NRTI that the patient has not taken for more than 14 days. In the case of lamivudine (3TC), naive means that the patient has never taken this drug.
* Are willing and able to drink 1.5 liters (a little over 1.5 quarts) of water or other fluids a day.
* Agree to use an effective barrier method of birth control (such as condoms) during the study and for 3 months after.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken protease inhibitors other than APV, NFV, SQV, or NFV plus SQV.
* Are resistant to the effects of IDV or RTV, as shown by a blood test. (Patients whose viral load is between 500 and 1,000 copies/ml will not need to be tested.)
* Have any active opportunistic (AIDS-related) infection in the 14 days before study entry.
* Have any medical condition or history of disease that would prevent them from completing the study or put them at risk.
* Have cancer that requires chemotherapy.
* Have an active infection that requires treatment in the 14 days before study entry.
* Have a fever for a week or more in the 30 days before study entry.
* Have taken nonnucleoside reverse transcriptase inhibitors (NNRTIs) in the 30 days before study entry.
* Have received a vaccine in the 21 days before study entry.
* Have received an experimental drug or a drug that affects the immune system in the 30 days before study entry.
* Have taken or plan to take certain other medications that may affect the study.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John G. Gerber, Study Chair; Edward P. Acosta, Study Chair
Locations (7):
- United States (7):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Acosta EP, Wu H, Hammer SM, Yu S, Kuritzkes DR, Walawander A, Eron JJ, Fichtenbaum CJ, Pettinelli C, Neath D, Ferguson E, Saah AJ, Gerber JG; Adult AIDS Clinical Trials Group 5055 Protocol Team. Comparison of two indinavir/ritonavir regimens in the treatment of HIV-infected individuals. J Acquir Immune Defic Syndr. 2004 Nov 1;37(3):1358-66. doi: 10.1097/00126334-200411010-00004. PMID 15483465
- [Result] King JR, Gerber JG, Fletcher CV, Bushman L, Acosta EP. Indinavir protein-free concentrations when used in indinavir/ritonavir combination therapy. AIDS. 2005 Jul 1;19(10):1059-63. doi: 10.1097/01.aids.0000174452.78497.54. PMID 15958837
- [Result] Wu H, Huang Y, Acosta EP, Park JG, Yu S, Rosenkranz SL, Kuritzkes DR, Eron JJ, Perelson AS, Gerber JG. Pharmacodynamics of antiretroviral agents in HIV-1 infected patients: using viral dynamic models that incorporate drug susceptibility and adherence. J Pharmacokinet Pharmacodyn. 2006 Aug;33(4):399-419. doi: 10.1007/s10928-006-9006-4. Epub 2006 Apr 1. PMID 16583266